CLINICAL TRIAL: NCT06121921
Title: A Pilot Study Assessing the Feasibility and Effectiveness of a Perioperative Multi-component Intervention in Patients With Acute Decompensated Aortic Stenosis Undergoing Urgent Transcatheter Aortic Valve Intervention
Brief Title: RESTORE-TAVI Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 330818
Record Dates: First submitted 2023-10-16; First posted 2023-11-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Frailty; Aortic Stenosis
MeSH Terms: conditions — Frailty; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Perioperative multi-component intervention
  Interventions: Other: Perioperative multi-component intervention
- Control (No Intervention): Routine inpatient care

INTERVENTIONS:
Other: Perioperative multi-component intervention — Physical Component
  Self-directed daily non-ambulatory exercise programme, comprising:
  * Rubber ball squeezes (3 sets of 12 reps, per hand)
  * Bicep curls (3 sets of 12 reps)
  * Leg extensions (3 sets of 12 reps)
  * Chair rises (3 sets of 12 reps)
  * Arm stretches (3 sets of 3 reps) Additional encouragement to mobilise
  Cognitive Component:
  Delirium prevention strategies including orientation, hydration, bowel/bladder function, infection control, analgesia, polypharmacy and cognitive stimulation
  Nutritional Component:
  * Formal dietician review if MUST score ≥ 2
  * IV ferritin if LVEF <45% and serum ferritin <100ng/mL or ferritin 100-299ng/mL with TSAT <20%
  Arms: Intervention

SUMMARY:
This is a pilot randomised control study assessing the feasibility and effectiveness of a perioperative multi-component intervention aimed at reducing adverse hospital events and improving functional outcomes in patients with acute decompensated aortic stenosis undergoing urgent transcatheter aortic valve implantation compared to standard care.

The intervention will consist of physical rehabilitation, delirium prevention, nutritional supplementation and anaemia correction (where indicated). The primary objective is to determine the feasibility and safety of delivering this intervention Secondary objectives include investigating the impact on adverse hospital events such as hospital-acquired disability and post-TAVI delirium, and on health-related quality of life and functional recovery following TAVI.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 70 years
2. Ability to provide written informed consent
3. Ability to speak English

Exclusion criteria:

1. Clinical instability defined as requiring use of inotropes/mechanical-circulatory support during admission or post-cardiac arrest
2. Active delirium (4AT score ≥ 4) at time of recruitment
3. Parkinson's disease (Hoehn & Yahr stage 3-5)
4. Recent stroke (within 7 days preceding recruitment)
5. Terminal condition (e.g. metastatic cancer) with life expectancy < 12 months
6. Clinical unsuitable for recruitment to trial according to the discretion of the research team

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment rates | 1 year
  Average number of patients per month willing to give informed consent and be randomised into a trial of a perioperative frailty intervention
Feasibility: Safety | On discharge: e.g. 2-7 days
  In-hospital adverse events (e.g. falls, ischaemia, arrhythmia, acute kidney injury), in-hospital mortality

SECONDARY OUTCOMES:
Incidence of hospital-acquired disability | 30 days
  defined as loss of ≥ 1 ADL at discharge compared to admission; and followed-up at 30 days after discharge
Incidence of delirium | Daily (during inpatient admission) until the seventh day post-TAVI and then twice weekly thereafter
  Assessed daily during hospitalisation by using 4AT until the seventh day post-TAVI and then twice weekly thereafter
Changes in health-related quality of life | 30 days
  Measured using EQ-5D-5L at baseline and 30 days post discharge via telephone
Changes in physical frailty | 30 days
  By comparing SARC-F (strength, assistance with walking, rise form a chair, climb stairs and falls) questionnaire at baseline and 30 days (via telephone) after discharge
Changes in physical frailty | On discharge: e.g. 2-7 days
  By comparing dominant handgrip strength at admission and discharge - average of 3 trials of maximal isometric grip measured in kilograms using a Jamar hydraulic hand dynamometer (Anatomy Supply Partners LLC, Georgia, USA).
Changes in physical frailty | On discharge: e.g. 2-7 days
  By comparing timed chair rises at admission and discharge - time (measures in seconds) to complete five chair rises without using arms.
Change in cognitive function | 30 days
  Assessed using T-MoCA at admission and 30 days post discharge via telephone
Change in mood | 30 days
  Assessed using HADS at admission and 30 days post discharge via telephone
Incidence of falls during hospitalisation | On discharge: e.g. 2-7 days
Length of hospital stay | On discharge: e.g. 2-7 days
  Duration of inpatient stay at tertiary centre
Discharge destination | On discharge: e.g. 2-7 days
  e.g. to patient's own home, long-term care facility or district general hospital
Unplanned readmissions | 30 days
  Measured at 30 days post discharge from tertiary centre using hospital records and patient telephone-interview
Mortality | 30 days
  Measured at 30 days post discharge using hospital records and NHS Spine database

CONTACTS AND LOCATIONS:
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No